CLINICAL TRIAL: NCT06051812
Title: A Prospective, Observational, Non-interventional, Single-center Study to Analyze the Relationship Between Proteinuria and Renal Perfusion in Renal Transplant Recipients
Brief Title: Proteinuria and Renal Perfusion in Renal Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: TxASL2020
Record Dates: First submitted 2023-07-10; First posted 2023-09-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pre-kidney Transplant; Living Donor Kidney Transplantation; Renal Perfusion; End Stage Renal Disease
Keywords: Kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease remains one of the major cause of mortality in renal transplant recipients, with the rate of cardiac death 10-times higher than that of the general population. An independent association between post-transplant proteinuria and cardiovascular risk has been previously reported. Diseased native kidneys with residual urine output or the transplanted kidney could be the source of proteinuria following renal transplantation. A clear differentiation of the source of proteinuria (native kidneys versus allograft) could be important for appropriate management.

Proteinuria from native kidneys falls rapidly after renal transplantation, and persistent or worsening proteinuria is usually indicative of allograft pathology. The mechanisms behind the resolution of proteinuria of native kidney origin in the early post-transplant period are not well described.

An association between vascular parameters of the macrocirculation and post-transplant proteinuria has been described. To the best of our knowledge no data is available describing a link between post-transplant proteinuria and vascular parameters of the microcirculation.

In this study our goal is to analyze in a clinical trial in patients with end stage renal disease and residual urine output the relationship between proteinuria and renal perfusion of native kidneys before and after renal transplantation. In addition the investigators analyse if pre or post-transplant proteinuria is associated vascular and circulatory changes in the retinal circulation.

Our hypothesis is that renal perfusion of native kidneys correlates with early post-transplant proteinuria. Moreover the investigators hypothesize that post-transplant proteinuria is associated with vascular remodeling processes of the microcirculation 2 and 4 to 12 months after transplantation. To prove this hypothesis the investigators aim to include 25 pre kidney transplant patients of our living donor kidney transplantation program.

Total duration of this study for each patient is 5-12 months with total 4 visits, of which all are performed at the Clinical Research Center of the Department of Nephrology and Hypertension, University of Erlangen-Nuremberg. This study is important to better understand the mechanisms behind the fall of proteinuria after renal transplantation and the association between post-transplant proteinuria and cardiovascular risk.

DETAILED DESCRIPTION:
Renal transplantation is the treatment of choice for patients with end-stage kidney disease. Although renal transplantation is associated with reduced morbidity and mortality compared to chronic dialysis, cardiovascular disease remains one of the major cause of mortality in this population, with the rate of cardiac death 10-times higher than that of the general population. Proteinuria is not only considered as a diagnostic marker of renal disease in both native as well as the transplanted kidney, but also is widely described as an independent risk factor for cardiovascular morbidity and mortality in general population. Analogous to its impact in the general population, an independent association between post-transplant proteinuria and cardiovascular risk has been previously reported. The prevalence of proteinuria in renal transplant recipients is reported between 10% and 45%. Fernandez-Fresnedo et al. demonstrated that persistent proteinuria doubles the risk of cardiovascular disease and all-cause mortality in renal transplant recipients. Diseased native kidneys with residual urine output or the transplanted kidney could be the source of proteinuria following renal transplantation. A clear differentiation of the source of proteinuria (native kidneys versus allograft) is important for appropriate management.

Proteinuria from native kidneys falls rapidly after renal transplantation, and persistent or worsening proteinuria is usually indicative of allograft pathology. The mechanisms behind the resolution of proteinuria of native kidney origin in the early post-transplant period are not well described. CNI-induced renal vasoconstriction causing reduction in urine output from the native kidneys may be an explanation for the early resolution of native kidney proteinuria. However, the resolution of proteinuria of native kidney origin post-transplant have been reported in the pre-cyclosporine era.

An association between vascular parameters of the macrocirculation and post-transplant proteinuria has been described. High-grade post-transplant proteinuria has been found to be associated with higher pulse wave velocity, which is a marker of arterial stiffness of large arteries. Up to our knowledge no data is available describing a link between post-transplant proteinuria and vascular parameters of the microcirculation. In this study our goal is to analyze in a clinical trial in patients with end stage renal disease and residual urine output the relationship between proteinuria and renal perfusion of native kidneys before and after renal transplantation. In addition the investigators analyse if pre- or post-transplant proteinuria is associated with vascular and circulatory changes in the retinal circulation.

This study is a single-centre clinical study with 25 pre-kidney transplant patients of our living donor kidney transplantation program. This is an exploratory and non-confirmatory study, in which the investigators analyse renal perfusion of native kidneys in patients with end stage renal disease before and after kidney transplantation. Our hypothesis is that renal perfusion of native kidneys correlates with early post-transplant proteinuria. Moreover the investigators hypothesize that post-transplant proteinuria is associated with vascular remodeling processes of the microcirculation 2 and 4-12 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 75 years
* Male and Female patients
* Patients evaluated and accepted for living donor kidney transplantation with residual urine output of at least 500 ml/24 hours
* Informed consent has to be given in written form

Exclusion Criteria:

* Patients in unstable conditions due to any kind of serious disease, that infers with the conduction of the trial
* active Drug or alcohol abuse
* Pregnant and breast-feeding patients
* Body mass index > 35 kg/m²
* Subjects who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V
* Implanted pacemakers or defibrillators
* Other implanted metallic devices, which are not MRI compatible
* Claustrophobia
* Any other relevant clinical contraindication of MRI examination

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be included in the study only if they satisfy all the inclusion criteria and are not precluded from participation by any of the exclusion criteria. 25 pre-kidney transplant patients of our living donar kidney transplantation program will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Perfusion of native kidneys measured by ASL-MRI | change from baseline perfusion of native kidneys at 2 months after renal transplantation
  The primary objective of the study is to analyze is to measure renal perfusion of native kidneys before and after renal transplantation

SECONDARY OUTCOMES:
Perfusion of transplant kidney measured by ASL-MRI | 2 months after renal transplantation
  analyze perfusion of renal transplant
Wall to lumen ratio of retinal arterioles by SLDF measurement | change from baseline Wall to lumen ratio of retinal arterioles at 2 months and 12 months after renal transplantation
  analyze wall to lumen ratio of retinal arterioles before and after renal transplant
Retinal capillary flow determined by SLDF measurement | change from baseline retinal capillary flow at 2 months and 12 months after renal transplantation
  analyze retinal capillary flow before and after renal transplant
Central systolic pressure assessed by Sphygmocor XCEL | change from baseline central systolic pressure at 2 months and 12 months after renal transplantation
  analyze central systolic pressure before and after renal transplant
Pulse pressure assessed by Sphygmocor XCEL | change from baseline pulse pressure at 2 months and 12 months after renal transplantation
  analyze pulse pressure before and after renal transplant
Pulse wave velocity assessed by Sphygmocor XCEL | change from baseline pulse wave velocity at 2 months and 12 months after renal transplantation
  analyze pulse wave velocity before and after renal transplant
estimated glomerular filtration rate assessed in our central lab | change from baseline estimated glomerular filtration rate at 2 months and 12 months after renal transplantation
  analyze estimated glomerular filtration rate before and after renal transplant
Cystatin C assessed in our central lab | change from baseline Cystatin C at 2 months and 12 months after renal transplantation
  analyze Cystatin C before and after renal transplant
Urinary albumin creatinine ratio assessed in our central lab | change from baseline urinary albumine creatinine ratio at 2 months and 12 months after renal transplantation
  analyze Urinary albumin creatinine ratio before and after renal transplant in both spot and 24-h urine

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Background] Ojo AO, Hanson JA, Wolfe RA, Leichtman AB, Agodoa LY, Port FK. Long-term survival in renal transplant recipients with graft function. Kidney Int. 2000 Jan;57(1):307-13. doi: 10.1046/j.1523-1755.2000.00816.x. PMID 10620213
- [Background] Liefeldt L, Budde K. Risk factors for cardiovascular disease in renal transplant recipients and strategies to minimize risk. Transpl Int. 2010 Dec;23(12):1191-204. doi: 10.1111/j.1432-2277.2010.01159.x. Epub 2010 Sep 7. PMID 21059108
- [Background] Chronic Kidney Disease Prognosis Consortium; Matsushita K, van der Velde M, Astor BC, Woodward M, Levey AS, de Jong PE, Coresh J, Gansevoort RT. Association of estimated glomerular filtration rate and albuminuria with all-cause and cardiovascular mortality in general population cohorts: a collaborative meta-analysis. Lancet. 2010 Jun 12;375(9731):2073-81. doi: 10.1016/S0140-6736(10)60674-5. Epub 2010 May 17. PMID 20483451
- [Background] Peterson JC, Adler S, Burkart JM, Greene T, Hebert LA, Hunsicker LG, King AJ, Klahr S, Massry SG, Seifter JL. Blood pressure control, proteinuria, and the progression of renal disease. The Modification of Diet in Renal Disease Study. Ann Intern Med. 1995 Nov 15;123(10):754-62. doi: 10.7326/0003-4819-123-10-199511150-00003. PMID 7574193
- [Background] Barnas U, Schmidt A, Haas M, Kaider A, Tillawi S, Wamser P, Mayer G. Parameters associated with chronic renal transplant failure. Nephrol Dial Transplant. 1997;12 Suppl 2:82-5. PMID 9269707
- [Background] Yildiz A, Erkoc R, Sever MS, Turkmen A, Ecder ST, Turk S, Kilicarslan I, Ark E. The prognostic importance of severity and type of post-transplant proteinuria. Clin Transplant. 1999 Jun;13(3):241-4. doi: 10.1034/j.1399-0012.1999.130304.x. PMID 10383104
- [Background] Fernandez-Fresnedo G, Escallada R, Rodrigo E, De Francisco AL, Cotorruelo JG, Sanz De Castro S, Zubimendi JA, Ruiz JC, Arias M. The risk of cardiovascular disease associated with proteinuria in renal transplant patients. Transplantation. 2002 Apr 27;73(8):1345-8. doi: 10.1097/00007890-200204270-00028. PMID 11981434
- [Background] Roodnat JI, Mulder PG, Rischen-Vos J, van Riemsdijk IC, van Gelder T, Zietse R, IJzermans JN, Weimar W. Proteinuria after renal transplantation affects not only graft survival but also patient survival. Transplantation. 2001 Aug 15;72(3):438-44. doi: 10.1097/00007890-200108150-00014. PMID 11502973
- [Background] Guliyev O, Sayin B, Uyar ME, Genctoy G, Sezer S, Bal Z, Demirci BG, Haberal M. High-grade proteinuria as a cardiovascular risk factor in renal transplant recipients. Transplant Proc. 2015 May;47(4):1170-3. doi: 10.1016/j.transproceed.2014.10.062. PMID 26036546
- [Background] D'Cunha PT, Parasuraman R, Venkat KK. Rapid resolution of proteinuria of native kidney origin following live donor renal transplantation. Am J Transplant. 2005 Feb;5(2):351-5. doi: 10.1111/j.1600-6143.2004.00665.x. PMID 15643995
- [Background] Laplante L, Beaudry C, Houde M. [Early disappearance of proteinuria attributed to the original kidneys after kidney transplantation]. Union Med Can. 1975 Feb;104(2):246-8. No abstract available. French. PMID 1099753
- See also: Homepage Clinical Research Center — https://www.medizin4.uk-erlangen.de/forschung/klinische-forschungsstation-crc/